CLINICAL TRIAL: NCT07145359
Title: Development and Evaluation of A Virtual Reality Intervention for Symptoms Management During Hematopoietic Stem Cell Transplantation
Brief Title: Virtual Reality Intervention for Symptom Management in Stem Cell Transplantation
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Halic University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2025/350-361
Record Dates: First submitted 2025-08-12; First posted 2025-08-28 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Cancer and / or Hematological Malignancy; Hematopoetic Stem Cell Transplantation; Nursing Interventions; Symptom Management; Virtual Reality; ALLOGENEIC HEMATOPOIETIC STEM CELL TRANSPLANTATION
MeSH Terms: conditions — Neoplasms; Hematologic Neoplasms

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): Participants in this group will receive standard clinical care during hematopoietic stem cell transplantation (HSCT) without any additional intervention. They will not be exposed to any virtual reality content during the procedure. This group serves as the comparator to evaluate the effects of the VR intervention.
- Experimental group (Experimental): Participants in this group will receive standard clinical care during hematopoietic stem cell transplantation (HSCT) along with a 15-minute virtual reality (VR) intervention. The VR intervention involves viewing a nature-themed immersive video through a Meta Quest 3 headset. Patients will select one of five pre-approved videos created or curated by the research team based on Attention Restoration Theory (ART). The VR session will begin one minute before the stem cell infusion and end at the 15th minute of the procedure. The intervention is administered under the supervision of the researcher.
  Interventions: Other: Virtual Reality Intervention

INTERVENTIONS:
Other: Virtual Reality Intervention — This intervention is distinguished by its integration of a structured, nurse-led virtual reality (VR) protocol specifically designed for symptom management during hematopoietic stem cell transplantation (HSCT). Unlike general VR distraction methods used in oncology, this intervention employs video content created by the research team in accordance with Attention Restoration Theory (ART), offering five preselected nature-themed options tailored to patient preferences. Prior to the procedure, eligible patients are introduced to the intervention one day in advance and given the opportunity to trial the VR equipment, ask questions, and select their preferred video. During the infusion, VR is initiated exactly one minute before the stem cell procedure and ends at the 15th minute, as recommended by the literature. Symptom assessments are conducted immediately before and after the intervention using validated tools, including the Distress Thermometer, State Anxiety Inventory, and the Edmonto
  Arms: Experimental group

SUMMARY:
The goal of this clinical trial is to evaluate whether a virtual reality (VR) intervention based on the Symptom Management Model can reduce physical and psychosocial symptoms during hematopoietic stem cell transplantation (HSCT) in adult patients undergoing allogeneic transplantation.

The main questions it aims to answer are:

Does the VR intervention reduce distress levels during HSCT?

Does the VR intervention decrease state anxiety and symptom severity compared to standard care?

Does the VR intervention positively affect physiological outcomes and engraftment times?

Researchers will compare a group receiving standard clinical care plus a VR nature-themed video during HSCT to a group receiving standard care only to see if the VR intervention improves symptom management outcomes.

Participants will:

Be randomly assigned to either the intervention or control group.

In the intervention group:

Watch a 15-minute nature-themed VR video during stem cell infusion using Meta Quest 3.

The video content will be specifically created by the research team based on the principles of Attention Restoration Theory (ART).

In both groups:

Complete pre- and post-intervention assessments including:

Distress Thermometer

State-Trait Anxiety Inventory

Edmonton Symptom Assessment Scale

Physiological measures (vital signs)

Engraftment tracking

Satisfaction and open-ended feedback forms

DETAILED DESCRIPTION:
This study is a randomized controlled pilot trial designed to evaluate the effectiveness of a virtual reality (VR) intervention, based on the Symptom Management Model (SYM), in managing physical and psychosocial symptoms during allogeneic hematopoietic stem cell transplantation (HSCT). The intervention is nurse-led and grounded in Attention Restoration Theory (ART), utilizing immersive 360° nature-themed videos created or selected by the research team. These videos are intended to support psychological relaxation, reduce distress, and shift patients' focus away from treatment-related discomfort.

Eligible participants will be adult patients scheduled for allogeneic HSCT using peripheral blood stem cells. Patients will be randomly assigned to either the intervention or control group using stratified block randomization. The intervention group will receive standard clinical care in addition to watching a 15-minute VR video during the stem cell infusion procedure, delivered via Meta Quest 3 headsets. The control group will receive standard care only.

One day before the HSCT procedure, the researcher will meet with the eligible patients to introduce the study, answer questions, and familiarize them with the VR equipment and video content. Patients in the intervention group will be allowed to choose one of five pre-approved nature-themed VR videos. On the day of transplantation, baseline data (distress, anxiety, symptoms, vitals) will be collected approximately 15 minutes before the procedure. The VR headset will be applied 3 minutes before the infusion begins, and the video will start 1 minute prior to the procedure. The infusion will proceed according to the institution's standard protocols. Vital signs will be recorded during the intervention by the researcher. Patients will be reminded that they can request to remove the headset at any point if they feel uncomfortable.

At the 15th minute of the HSCT infusion, the video will end. Post-intervention assessments will include distress, anxiety, symptom severity, and satisfaction. If the patient does not feel well enough immediately after the session, additional time will be provided before collecting post-test data. To prevent infection risks, VR equipment will be disinfected after each use.

In addition to psychological and symptomatic outcomes, physiological parameters (blood pressure, heart rate, body temperature, oxygen saturation, respiratory rate) will be tracked. Neutrophil and platelet engraftment status will be assessed on Day +28 post-transplant. Patient satisfaction with the intervention will be measured using a visual analog scale and open-ended feedback.

This is the first known Turkish study to implement a theory-based, nurse-led virtual reality intervention during HSCT with the goal of symptom management. It is expected to provide valuable insight into the integration of digital care tools in supportive oncology nursing practice.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years or older
* Able to speak and understand Turkish
* Scheduled to undergo allogeneic hematopoietic stem cell transplantation (HSCT)
* Receiving stem cell products collected from peripheral blood
* Voluntarily agree to participate in the study and provide informed consent

Exclusion Criteria:

* Undergoing autologous hematopoietic stem cell transplantation
* Receiving stem cell products collected from bone marrow
* Diagnosed with medical or psychiatric comorbidities that could interfere with participation, as reported by the healthcare team
* Presenting infection symptoms (e.g., respiratory, gastrointestinal) that may contaminate study equipment, as identified by the healthcare team
* Having visual, auditory, verbal, or cognitive impairments that may prevent interaction with the VR equipment
* Previously received any form of hematopoietic stem cell transplantation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-09-10 (Estimated); Primary Completion 2026-06-10 (Estimated); Study Completion 2026-09-10 (Estimated)

PRIMARY OUTCOMES:
Change in Distress Level | From 15 minutes before HSCT infusion to 15 minutes after the start of infusion
  Assessed using the Distress Thermometer. Scores range from 0 (no distress) to 10 (extreme distress).
Change in State Anxiety | From 15 minutes before HSCT infusion to 15 minutes after the start of infusion
  Assessed using the State subscale of the State-Trait Anxiety Inventory (STAI).
Change in Symptom Severity | 15 minutes before HSCT infusion to 15 minutes after the start of infusion
  Evaluated using the Edmonton Symptom Assessment Scale (ESAS) including pain, fatigue, nausea, depression, anxiety, appetite loss, dyspnea, sleep disturbance, and overall well-being.

SECONDARY OUTCOMES:
Change in Systolic Blood Pressure | Baseline (pre-HSCT infusion), during HSCT infusion, and immediately post-infusion (within 30 minutes)
  Change in systolic blood pressure (mmHg)
Change in Diastolic Blood Pressure | Baseline (pre-HSCT infusion), during HSCT infusion, and immediately post-infusion (within 30 minutes)
  Change in diastolic blood pressure (mmHg)
Change in Heart Rate | Baseline (pre-HSCT infusion), during HSCT infusion, and immediately post-infusion (within 30 minutes)
  Change in heart rate (beats per minute)
Change in Body Temperature | Baseline (pre-HSCT infusion), during HSCT infusion, and immediately post-infusion (within 30 minutes)
  Change in body temperature (°C)
Change in Oxygen Saturation | Baseline (pre-HSCT infusion), during HSCT infusion, and immediately post-infusion (within 30 minutes)
  Change in oxygen saturation (%)
Change in Respiratory Rate | Baseline (pre-HSCT infusion), during HSCT infusion, and immediately post-infusion (within 30 minutes)
  Change in respiratory rate (breaths per minute)
Neutrophil Engraftment Time | Assessed on Day +28 post-transplant
  Defined as the number of days from HSCT to the first of three consecutive days with absolute neutrophil count ≥500/mm³
Platelet Engraftment Time | Assessed on Day +28 post-transplant
  Defined as the number of days from HSCT to the first of three consecutive days with platelet count ≥20,000/mm³ without transfusion
Patient Satisfaction (Visual Analog Scale) | Within 15 minutes after HSCT infusion
  Patient satisfaction will be assessed using the Visual Analog Scale (VAS; range 0-10 cm), where 0 = not satisfied at all (worst outcome) and 10 = extremely satisfied (best outcome). Higher scores indicate greater patient satisfaction.
Patient Satisfaction (Qualitative Feedback Form) | Within 15 minutes after HSCT infusion
  Patient satisfaction with the virtual reality experience will be assessed using an open-ended feedback form. Patients will be invited to provide narrative responses addressing the following aspects:
  Whether they were satisfied with the VR experience, Any side effects experienced (e.g., dizziness, nausea, discomfort), Suggestions for improvement.

IPD SHARING:
Plan to Share IPD: No